CLINICAL TRIAL: NCT06965088
Title: Comparison of Recurrence Rate of Keloid After Excision Between Intra-operative Steroid Injection and Steroid With Platelet-rich Plasma Injection Combination Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Chanokchon Kongkergkiat, Chanokchon Kongkergkiat, M.D., Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2024/502
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Patients With Keloid Scar
Keywords: Keloid; Steroid; Triamcinolone; Platelet rich plasma; PRP
MeSH Terms: conditions — Keloid | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-operative corticosteroid injection (Active Comparator): Intra-operative corticosteroid injection alone was administered around the surgical wound using triamcinolone acetonide (40 mg/ml). The injection was performed into the intradermal layer using a 30G needle, immediately after keloid excision and wound closure. The medication was injected along the wound edges following the suture line, at a dosage of 0.1 ml per 1 centimeter of wound length.
  Interventions: Drug: Intra-operative corticosteroid injection
- Combined Intra-operative platelet-rich plasma with corticosteroid injection (Experimental): Combined Intra-operative platelet-rich plasma with corticosteroid injection was administered around the surgical wound. Each patient had 10 ml of blood collected into a RegenKit A-PRP tube. The blood-filled tube was then placed into a RegenLab PRP centrifuge and spun for approximately 5 minutes to obtain platelet-rich plasma (PRP), yielding around 5 ml of injectable PRP. Once prepared, the PRP was stored in the collection tube and used within 4 hours from the time of blood draw to the time of injection. After the keloid excision and wound closure were completed, the PRP was aseptically aspirated from the tube using a sterile needle and injected into the intradermal layer along the wound edges using a 30G needle. The injection was performed in a sterile manner, with a dosage of 0.5 ml of PRP per 1 centimeter of wound length. For corticosteroid administration, triamcinolone acetonide (40 mg/ml) was used. The medication was injected into the intradermal layer using a 30G needle along the
  Interventions: Biological: Combined Intra-operative platelet-rich plasma with corticosteroid injection

INTERVENTIONS:
Biological: Combined Intra-operative platelet-rich plasma with corticosteroid injection — Combined Intra-operative platelet-rich plasma with corticosteroid injection was administered around the surgical wound. Each patient had 10 ml of blood collected into a RegenKit A-PRP tube. The blood-filled tube was then placed into a RegenLab PRP centrifuge and spun for approximately 5 minutes to obtain platelet-rich plasma (PRP), yielding around 5 ml of injectable PRP. Once prepared, the PRP was stored in the collection tube and used within 4 hours from the time of blood draw to the time of injection. After the keloid excision and wound closure were completed, the PRP was aseptically aspirated from the tube using a sterile needle and injected into the intradermal layer along the wound edges using a 30G needle. The injection was performed in a sterile manner, with a dosage of 0.5 ml of PRP per 1 centimeter of wound length. For corticosteroid administration, triamcinolone acetonide (40 mg/ml) was used. The medication was injected into the intradermal layer using a 30G needle along the
  Arms: Combined Intra-operative platelet-rich plasma with corticosteroid injection
Drug: Intra-operative corticosteroid injection — Intra-operative corticosteroid injection alone was administered around the surgical wound using triamcinolone acetonide (40 mg/ml). The injection was performed into the intradermal layer using a 30G needle, immediately after keloid excision and wound closure. The medication was injected along the wound edges following the suture line, at a dosage of 0.1 ml per 1 centimeter of wound length.
  Arms: Intra-operative corticosteroid injection

SUMMARY:
Keloid scars are benign skin lesions characterized by excessive collagen deposition, and their treatment remains challenging due to a high recurrence rate even after surgical excision. Combination therapies have been shown to be more effective than monotherapy. A common approach for treating recurrent keloids is surgical excision followed by intralesional corticosteroid injection; however, recurrence rates remain substantial. This study was conducted to evaluate the recurrence rate of keloid scars following surgical excision combined with intralesional corticosteroid and platelet-rich plasma (PRP) injection, compared to corticosteroid injection alone administered intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Having keloid scars less than 10 centimeters in length
* Undergoing complete keloid excision (extralesional excision)
* Undergoing surgery under local anesthesia

Exclusion Criteria:

* Patients currently receiving immunosuppressive drugs or systemic steroids
* Patients with chronic diseases under active treatment, such as tuberculosis
* Pregnant or breastfeeding women
* Patients likely to have poor treatment adherence, such as those with cancer, epilepsy, or psychiatric disorders
* Patients with vascular diseases or hematologic/coagulation abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of keloid | Within 12 months after end of the intervention
  Vancouver scar scale

SECONDARY OUTCOMES:
Itching at scar | Within 12 months after end of the intervention
  Patient reported outcome using a questionnaire interview
Pain at scar | Within 12 months after end of the intervention
  Patient reported outcome using a questionnaire interview
Skin atrophy | Within 12 months after end of the intervention
  Clinical examination
Skin telangiectasia | Within 12 months after end of the intervention
  Clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided